CLINICAL TRIAL: NCT03290170
Title: Radiostereometric Analysis of Gap Balancing Versus Measured Resection for the Journey II Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Douglas Naudie, Orthopaedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109512
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Knee Osteoarthritis; Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measured resection technique (Experimental): Measured resection surgical technique
  Interventions: Procedure: Measured Resection
- Gap Balancing Technique (Experimental): Gap Balancing surgical technique
  Interventions: Procedure: Gap Balancing

INTERVENTIONS:
Procedure: Measured Resection — Bony landmarks are used to set femoral component rotation.
  Arms: Measured resection technique
Procedure: Gap Balancing — Relies on ligament releases prior to bone cuts.
  Arms: Gap Balancing Technique

SUMMARY:
This is a randomized study comparing the measured resection and gap-balancing surgical techniques for total knee replacement (TKR) using a cemented Journey II TKR implant system. We will be comparing the two surgical methods by evaluating implant migration using radiostereometric analysis (RSA) imaging, evaluating contact kinematics (knee mechanics) through RSA under dynamic conditions and comparing patient knee outcome scores.

DETAILED DESCRIPTION:
The stability of a total knee replacement (TKR) surgery depends on soft tissue balance (i.e. balance of supporting ligaments) and bony cuts made during surgery that dictate the rotation of the femoral (thigh bone) component. Two main techniques predominate for execution of the bone cuts and soft tissue balance in TKR. In measured resection, pre-determined bony cuts are made and appropriate balance is obtained by judicious soft tissue releases as required. In gap balancing, the bony cuts for femoral rotation are driven by the native soft tissues. How these two surgical approaches affects the biomechanics of the knee invivo is unclear. The purpose of this study is to examine the patello-femoral articulation as well as coronal balance of the respective techniques under dynamic conditions. Secondary goals will be to examine the impact on femoral component position on changes to coronal plane position through a range of flexion/extension. As patellofemoral symptoms and flexion instability are two of the most common causes of patient dissatisfaction and revision in the short term, this study has the potential to have significant patient impact. The study also has the potential to provide information on long term wear potential if articular incongruity is found. TKA is a procedure that has good results in most patients, however, up to 20% of patients are not satisfied with their outcome. (1) Some of these dissatisfied patients require early revision. Early revisions are often attributed to technical issues, such as revisions required for instability, patellofemoral symptoms, stiffness or aseptic loosening (2). This highlights the impact of surgical technique on clinical outcomes. There are two main philosophies on how to complete bone resections and achieve a balanced TKA. The measured resection technique utilizes a standard set of bony cuts based on bony landmarks and then balances the knee by making judicious soft tissue releases. Component position, particularly femoral rotation, is fairly constant with using this technique. Gap balancing adjusts the bony cuts for femoral rotation to balance the soft tissues of the knee in flexion, potentially avoiding the necessity of soft tissue releases. In contrast to the measured resection technique, gap balancing allows for variable rotation of the femoral component. This variability in femoral rotation has the potential to impacts the coronal plane motion as well as tracking at the patellofemoral articulation. Surgeons have strong opinions that both the gap balanced (3) and measured resection techniques (4) provide superior results. However, in spite of a variety of literature in support of each technique, little has been done to compare the biomechanics of each technique. There is a lack of scientifically rigorous assessment of the impact of surgical technique on femoral rotation, with resultant changes to coronal plane motion. This prevents the elucidation of potential sources of clinical outcome differences both in the short term and the long term. The impact of femoral component rotation will be examined by examining the coronal plane motion. An area impacted by the two TKA techniques is how they impact coronal plane motion in flexion. There has only been one paper written utilizing dynamic fluoroscopy to examine the differences in techniques (7). This study examined lift-off of the lateral component in a comparative study of the two techniques using dynamic fluoroscopy. This study was limited in nature, with only the ability to quantify the amount of separation of the femoral component from the tibial component in flexion. It did not examine the impact of femoral rotation on flexion alignment, or correlate patient satisfaction scores to the dynamic fluoroscopy findings. With the combination of advanced imaging to determine component position with respect to bony landmarks (8) as well as dynamic fluoroscopy, a large area of new information can be gathered. Examination of the impact of surgical technique with the use of cement to femoral component rotation, and how this impacts coronal plane motion are achievable goals, with potential for a significant impact on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* Primary, unilateral total knee arthroplasty

Exclusion Criteria:

* History of alcoholism
* Inability to speak or read English (questionnaires are only provided in English)
* Pregnant women and women with plans to begin a family
* Inflammatory arthritis -Bilateral total knee arthroplasty
* Revision total knee arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Implant migration | 2 and 6 weeks, 3, 6 and 12 months and 2 years post-operatively
  Comparison of the two surgical techniques using radiostereometric analysis (RSA) imaging

SECONDARY OUTCOMES:
Contact Kinematics Under Dynamic Conditions | 3 and 12 months post-operatively
  Comparison of the two surgical techniques using radiostereometric analysis (RSA) imaging

OTHER OUTCOMES:
Patient-reported outcomes (PROs) | 2 and 6 weeks, 3, 6 and 12 months and 2 years post-operatively
  Comparison of the two surgical techniques using PROs

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Naudie, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada